CLINICAL TRIAL: NCT05876312
Title: A Phase 1, Randomized, Double Blind, Placebo-Controlled, Single Ascending Dose Study in Healthy Participants Followed by a Phase 2a Open Label Study in Participants With PNH and Residual Anemia to Evaluate the Safety, Tolerability, PK and PD of ADX-038
Brief Title: Safety, Tolerability, PK and PD of ADX-038 in Healthy Participants and Paroxysmal Nocturnal Hemoglobinuria (PNH) Patients
Acronym: PNH
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ADARx Pharmaceuticals, Inc. (Industry)
Collaborators: ADARx Australia Pty Ltd (Unknown); Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ADX-038-101
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria (PNH)
Keywords: siRNA; PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal | interventions — RNA, Small Interfering; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Participant, Care Provider, Investigator
Masking Description: Masking is only applicable to Phase 1 in HP. Phase 2a is open label and there is no masking.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Phase 1 - Active ADX-038 administered to HP (Experimental): For each cohort in Phase 1 (SAD), 8 participants will be randomized in a 3:1 ratio; 6 participants to active (ADX-038): 2 participants to control (matched placebo). Randomization will be on Day 1. Initially, 2 sentinel participants (1 active and 1 placebo) will be randomized and dosed. The sentinel participants will be evaluated for safety. The investigator's assessment and the independent medical monitor will decide upon the randomization and dosing of the 6 remaining participants (5 active and 1 placebo) according to the randomization schedule.
  Interventions: Drug: ADX-038
- Phase 1- Placebo administered to HP (Placebo Comparator): For each cohort in Phase 1 (SAD), 8 participants will be randomized in a 3:1 ratio; 6 participants to active (ADX-038): 2 participants to control (matched placebo). Randomization will be on Day 1. Initially, 2 sentinel participants (1 active and 1 placebo) will be randomized and dosed. The sentinel participants will be evaluated for safety. The investigator's assessment and the independent medical monitor will decide upon the randomization and dosing of the 6 remaining participants (5 active and 1 placebo) according to the randomization schedule.
  Interventions: Drug: Placebo
- Phase 2a - ADX-038 administered to PNH participants (Experimental): This will be initiated at the dose level determined by the Safety Review Committee from SAD in HPs. The treatment of PNH participants is an open-label study.
  Interventions: Drug: ADX-038

INTERVENTIONS:
Drug: ADX-038 — siRNA duplex oligonucleotide
  Other Names: siRNA
  Arms: Phase 1 - Active ADX-038 administered to HP; Phase 2a - ADX-038 administered to PNH participants
Drug: Placebo — Saline
  Other Names: Saline
  Arms: Phase 1- Placebo administered to HP

SUMMARY:
The first-in-human Phase 1/Phase 2a study described herein will evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics (PD) of ADX-038 in both healthy participants (HP) and in patients with paroxysmal nocturnal hemoglobinuria (PNH).

DETAILED DESCRIPTION:
The clinical study described in this protocol is a Phase 1/Phase 2a study evaluating safety, tolerability, PK, and PD of ADX-038.

The study consists of 2 parts:

1. Phase 1 - Randomized, double-blind, placebo-controlled, parallel group, single ascending dose (SAD) in HP with up to 5 dose cohorts.
2. Phase 2a - Open label, single-arm (ADX-038), 2 dose study in participants with paroxysmal nocturnal hemoglobinuria (PNH) and residual anemia on a standard-of-care (SOC) anti-C5 regimen of ravulizumab or eculizumab.

ELIGIBILITY:
Phase 1 Key Inclusion Criteria

* 18 to 55 years of age
* Participants who are healthy as determined by medical evaluation
* History of recent meningococcal, pneumococcal and Haemophilus influenzae type B vaccinations or willing to be vaccinated
* Screening tests negative for illicit drug, nicotine, and alcohol use

Phase 1 Key Exclusion Criteria

* History of any significant medical conditions, except for completely excised non-melanoma skin cancer or low grade cervical intraepithelial neoplasia without evidence of recurrence within the prior 3 months
* Any viral, bacterial, parasitic, or fungal infection within the prior 30 days
* Frequent respiratory, nasopharyngeal or ear infections (more than 5 infections per year)
* History of environmental exposure or sick contact that increase the risk of meningococcal, pneumococcal and/or Haemophilus influenza type B infections
* Complement deficiency or immunodeficiency syndrome
* Major surgery or significant traumatic injury within the prior 3 months
* History of anaphylaxis or hypersensitivity reactions
* History of penicillin allergy
* History of splenectomy
* History of alcohol abuse or illicit drug use
* Donated plasma within the prior 7 days
* Donated blood or loss more than 400 milliliters of blood (excluding blood volume drawn at screening) within the prior 90 days
* Screening estimated creatinine clearance of less than 60 milliliters per minute
* Screening hematology, serum chemistry, or coagulation parameters that are outside the normal range
* Screening vital signs that are abnormal per protocol specification
* Screening electrocardiogram findings that are clinically significant
* Pregnant or lactating females
* Use of prescription (except for contraceptives and study-related prophylactic antibiotics) or over-the counter medications (except for paracetamol or ibuprofen) or vitamins/supplements within the prior 7 days
* Use of medications that may reduce the effectiveness of hormonal contraceptives within the prior 28 days
* Use of an investigational therapeutics within the prior 30 days or within the expected washout (at least 5 half-lives)
* Unwilling or unable to adhere to study-related prophylactic antibiotics requirements

Phase 2a Key Inclusion Criteria

* at least 18 years of age
* Diagnosis of paroxysmal nocturnal hemoglobinuria based on documented clone size
* Hemoglobin concentration of less than 12 gram per deciliter
* History of recent meningococcal, pneumococcal and Haemophilus influenzae type b vaccinations or willing to be vaccinated
* On a stable anti-C5 regimen for greater than or equal to 12 weeks prior to Day 1

Phase 2a Key Exclusion Criteria

* Any viral, bacterial, parasitic, or fungal infection within the prior 14 days
* HIV, active hepatitis C or hepatitis B infection
* History of meningococcal or tuberculosis infection
* History of malignancy in the past 5 years, except for completely excised non-melanoma skin cancer or low grade cervical intraepithelial neoplasia with no evidence of recurrence within the prior 3 months
* Complement deficiency syndrome
* History of hematopoietic stem cell transplantation
* History of splenectomy
* Inflammatory bowel disease, systemic lupus erythematosus, rheumatoid arthritis, or chronic liver disease
* Clinically significant and uncontrolled medical conditions including, but not limited to, thromboembolic disease, acute coronary syndrome, and diabetes
* Pregnant or lactating females
* Use of an investigational therapeutics within the prior 30 days or within the expected washout period (at lest 5 half-lives)
* Abstain from alcohol consumption for 48 hrs before day of dosing and restrict to no more than an average of 14 standard drinks per week

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety in Healthy Volunteers | 365 days
  To evaluate the safety and tolerability of ADX-038 in HVs by incidence, relationship, and severity of adverse events and serious adverse events
Safety in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Evaluate the safety and tolerability of ADX-038 by incidence, relationship, and treatment-emergent adverse events and serious adverse events.

SECONDARY OUTCOMES:
Pharmacokinetics in Healthy Participants | 8 days
  To characterize the Pharmacokinetics of ADX-038 in HPs by measuring the Maximum observed plasma concentration (Cmax)
Pharmacodynamics in Healthy Participants | 365 days
  Change from base in plasma concentrations over time in Complement factor B (CFB) protein via assay measurement
Pharmacodynamics in Paraxysmal Nocturnal Hemoglobinuria | 365 days
  Evaluate the changes in hemoglobin concentrations
Pharmacodynamics in Paraxysmal Nocturnal Hemoglobinuria | 365 days
  Characterize the changes in serum concentration of complement factor B (CFB) protein and complement alternative pathway activity level.
Pharmacodynamics in Healthy Participants | 365 days
  Change in complement alternative pathway activity via assay measurement

OTHER OUTCOMES:
Immune Response in Healthy Participants | 365 days
  Anti-polyethylene glycol (PEG) antibody titers and anti-drug antibody titers
Pharmacodynamics in Healthy Participants | 365 days
  Change in complement classical pathway activity via assay measurement
Safety in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Evaluate the change from baseline in follow up visits for safety assesments
Clinical Effect in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Look at time (number of days) from dosing (Day 1) to diminished therapeutics effect (DTE)
Efficacy in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Evaluate changes in lactate dehydrogenase (LDH) (U/L)
Effects on Hemolysis in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Evaluate incidence of clinical breakthrough hemolysis, blood transfusions and Incidence of major adverse vascular events (MAVEs)
Pharmacokinetics in Paraxysmal Nocturnal Hemoglobinuria | 8 days
  Characterize PK parameters of ADX-038 by plasma C(max)
Pharmacodynamics in Paraxysmal Nocturnal Hemoglobinuria | 365 days
  Characterize changes in complement classical pathway activity level
Immune Response in Paraxysmal Nocturnal Hemoglobinuria | 365 days
  Determine Anti-PEG and anti-drug antibody titers
Efficacy in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Evaluate changes in serum free hemoglobin
Efficacy in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Evaluate changes in Haptoglobin Concentrations
Efficacy in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Evaluate changes in Reticulocyte Counts (%)
Efficacy in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Evaluate changes in Bilirubin (umol/L)
Efficacy in Paroxysmal Nocturnal Hemoglobinuria Participants | 365 days
  Evaluate changes in Aspartate aminotransferase (U/L)
Pharmacokinetics in Paraxysmal Nocturnal Hemoglobinuria | 8 days
  Characterize PK parameters of ADX-038 by plasma AUC (0-infinity)
Pharmacokinetics in Paraxysmal Nocturnal Hemoglobinuria | 8 days
  Characterize PK parameters of ADX-038 by plasma AUC(0-last)
Pharmacokinetics in Paraxysmal Nocturnal Hemoglobinuria | 8 days
  Characterize PK parameters of ADX-038 by plasma T(max)

CONTACTS AND LOCATIONS:
Locations (4):
- Australia (3):
  - Nucleus Network Brisbane, Brisbane, Queensland
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
- Richmond Pharmacology Ltd, London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No